CLINICAL TRIAL: NCT05706350
Title: Evaluating the Effect of Different Daily Plant Stanol Ester Intakes on the Vaccination Response to an Influenza Vaccine
Brief Title: Plant Stanol Esters and Influenza Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Raisio Nutrition Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 22-048
Record Dates: First submitted 2023-01-11; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Immune Response
Keywords: Plant Stanols; Immune system; Influenza vaccination
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Plant stanol group (2 grams per day) (Experimental): Dietary Supplement: 4 soft chews containing 0.5g plant stanols each (delivered as plant stanol esters) Soft chews containing 0.5g plant stanols each delivered as plant stanol esters
  Interventions: Biological: Influenza vaccine; Dietary Supplement: Plant stanol soft chews (2g per day)
- Plant stanol group (3 grams per day) (Experimental): Dietary Supplement: 6 soft chews containing 0.5g plant stanols each (delivered as plant stanol esters) Soft chews containing 0.5g plant stanols each delivered as plant stanol esters
  Interventions: Biological: Influenza vaccine; Dietary Supplement: Plant stanol soft chews (3g per day)
- Plant stanol group (4 grams per day) (Experimental): Dietary Supplement: 8 soft chews containing 0.5g plant stanols each (delivered as plant stanol esters) Soft chews containing 0.5g plant stanols each delivered as plant stanol esters
  Interventions: Biological: Influenza vaccine; Dietary Supplement: Plant stanol soft chews (4g per day)
- Placebo group (Placebo Comparator): Dietary Supplement: 6 placebo soft chews Soft chews that do not contain plant stanols
  Interventions: Biological: Influenza vaccine; Dietary Supplement: Control soft chews

INTERVENTIONS:
Biological: Influenza vaccine — Single dose of the Influenza vaccine Participants have to wait until they are invited to receive the vaccine by the general practitioner; this study does not interfere with national planning of the vaccine
Dietary Supplement: Plant stanol soft chews (2g per day) — Participants have to consume 4 soft chews per day containing 0.5g plant stanols each (delivered as plant stanol esters), corresponding to a total plant stanol intake of 2g daily
  Arms: Plant stanol group (2 grams per day)
Dietary Supplement: Plant stanol soft chews (3g per day) — Participants have to consume 6 soft chews per day containing 0.5g plant stanols each (delivered as plant stanol esters), corresponding to a total plant stanol intake of 3g daily
  Arms: Plant stanol group (3 grams per day)
Dietary Supplement: Plant stanol soft chews (4g per day) — Participants have to consume 8 soft chews per day containing 0.5g plant stanols each (delivered as plant stanol esters), corresponding to a total plant stanol intake of 4g daily
  Arms: Plant stanol group (4 grams per day)
Dietary Supplement: Control soft chews — Participants have to consume 6 control soft chews per day that does not contain plant stanols
  Arms: Placebo group

SUMMARY:
Plant stanols are known to lower low-density lipoprotein cholesterol (LDL-C). However, recent studies have suggested that these compounds also beneficially influence the immune system, e.g. increasing vaccine-specific antibody titers. BMI and age have previously been negatively associated to vaccination responses. If plant stanols indeed have beneficial effects on the immune system, people with overweight or obesity and higher age might benefit from consuming plant stanols prior to receiving the influenza vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 60 years or older (or 59, but turning 60 years during influenza season 2022/2023 (in line with RIVM guidelines))
* BMI between 20 and 35 kg/m2
* Currently not using products containing plant sterols or stanols (products with a cholesterol lowering claim of Becel ProActiv, Benecol, Danacol, store brands)
* Willing to abstain from products containing plant sterols or stanols during the study (products with a cholesterol lowering claim of Becel ProActiv, Benecol, Danacol, store brands)
* Willing to keep the intake of fish oil and vitamin supplements constant

Exclusion Criteria:

* Already received influenza vaccination in 2022
* Already had influenza in 2022
* Allergy to an ingredient of the chews
* Having donated blood within one month prior to the start of the study, or planning to donate blood during the study
* Excessive alcohol use (>20 consumptions per week)
* Regular use of soft and/or hard drugs

Min Age: 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Vaccine specific IgM antibody titer | Maximal change from T=0 (change T=0 to T=3 weeks or T=4 weeks)
  The response to the Influenza vaccine will be measured by quantifying the specific IgM antibody titer

SECONDARY OUTCOMES:
Vaccine specific IgG antibody titer | T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  The response to the Influenza vaccine will be measured by quantifying the specific IgG antibody titer
Immune parameters (1) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Cytokine production by PBMCs after stimulation with antiCD3-antiCD28 antiCD28 antibodies using the TruCulture system
Immune parameters (2) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  hsCRP
Leukocyte count | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Number of leukocytes measured in EDTA plasma
Leukocyte differential count | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Number of subgroups of leukocytes measured in EDTA plasma
Fasted metabolism (1) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Serum non-cholesterol sterols and stanols
Fasted metabolism (2) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Serum lipid and lipoprotein profile
Fasted metabolism (3) | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Plasma glucose
Anthropometry (1) | Day - 1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Body weight
Anthropometry (2) | Day - 1 (start study)
  Height
Anthropometry (3) | Day - 1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Waist circumference
Anthropometry (4) | Day - 1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Hip circumference
Anthropometry (5) | Day - 1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Waist-to-hip ratio
Diet | Day - 1 (start study), T=4 weeks after vaccination (end of study)
  Food frequency questionnaire is used to determine if the participants maintain their habitual diet and to determine if the participants do not consume plant stanols and/or sterols outside the intervention
Liver elastography | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Fibroscan
Liver fat content | Day - 1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination (end of study)
  Fibroscan
Diary outcomes (1) | Day - 1 (start study), T=4 weeks after vaccination (end of study)
  Adverse events as assessed by the diary
Diary outcomes (2) | Day - 1 (start study), T=4 weeks after vaccination (end of study)
  Medication intake as assessed by the diary

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands